CLINICAL TRIAL: NCT03046537
Title: Detection of PCOS and Ovulation Timing by NA-Nose
Brief Title: Detection of PCOS by Sensors Array
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 020916COM1k
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Metabolic State, Breath Analysis, NA-Nose
MeSH Terms: interventions — Breath Tests

STUDY DESIGN:
Intervention Model Description: ovulatory women will be compared to women who do not ovulate regularly (PCOS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ovulatory (Active Comparator): Comparison in metabolic state between ovulatory and PCOS women by collecting breath test from participant.
  Interventions: Diagnostic Test: Breath test
- PCOS (Active Comparator): Comparison in metabolic state between ovulatory and PCOS women by collecting breath test from participant
  Interventions: Diagnostic Test: Breath test

INTERVENTIONS:
Diagnostic Test: Breath test — Collecting breath test from participants

SUMMARY:
Detection of metabolic state of women with polycystic ovary using NA-Nose.

DETAILED DESCRIPTION:
Breath of women undergoing fertility treatment including PCOS and ovulatory women will be collected and transferred for our labs for further analysis in define the metabolic state. The detection will be made using sensors arrays and GCMS.

ELIGIBILITY:
Inclusion Criteria:women undergoing follow up for ovulation detection. -

Exclusion Criteria:Pregnancy

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Detection of different metabolic state between groups. | two years
  Finding that there special markers in the breath test that indicate a different metabolic state in PCOS.

IPD SHARING:
Plan to Share IPD: No